CLINICAL TRIAL: NCT04528472
Title: Longhua Hospital, Shanghai University of TCM
Brief Title: Acute Ischemic Apoplexy Syndrome Specificity and Acupuncture Intervention Research
Acronym: AIAI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: longhuaacup
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Acute Ischemia
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Treatment (Experimental): Acupuncture Treatment: main point: DU20, DU24, MS7, LI4, ST40 Oral Medicine Rehabilitation Treatment
  Interventions: Other: Acupuncture Treatment
- Regular Treatment (Experimental): Acupuncture Treatment Oral Medicine Rehabilitation Treatment
  Interventions: Other: Regular Treatment

INTERVENTIONS:
Other: Acupuncture Treatment — stimulate acupoints to accelerate recovery
  Arms: Acupuncture Treatment
Other: Regular Treatment — Oral Medicine and Rehabilitation Treatment
  Arms: Regular Treatment

SUMMARY:
This project optimizes the TCM Symptoms and Symptoms Scale. A curative effect evaluation system of acupuncture in the treatment of acute ischemic stroke is formed to provide clinical evidence by the following indexes: neurological impairment, motor dysfunction, TCM Symptoms and Symptoms Scale, combined with the patients' head MRI, Plasma BDNF, MMP-9 and other biomarkers.

DETAILED DESCRIPTION:
Based on the previous work, this project optimizes the TCM Symptoms and Symptoms Scale. Through the cohort study method, 194 patients with acute ischemic stroke were evaluated for neurological impairment, motor dysfunction, TCM Symptoms and Symptoms Scale, combined with the patients' head MRI. , Plasma BDNF, MMP-9 and other biomarkers, screen TCM syndromes related to stroke outcome indicators, and adopt targeted comprehensive acupuncture and moxibustion program intervention and follow-up to establish a stroke-specific intervention outcome prediction model with TCM characteristics. A curative effect evaluation system of acupuncture and moxibustion in the treatment of acute ischemic stroke is formed to provide clinical evidence.

ELIGIBILITY:
Inclusion Criteria:

* (1) It meets the diagnostic criteria in the "Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2014"; with the support of brain CT or MRI imaging examination, the vital signs are stable, the state of consciousness is clear, and the GCS>8 points; （2）.Onset is less than 2 weeks; （3）. There is no indication for thrombolysis, or the patient do not accept thrombolysis; （4）. For moderate to severe patients, the National Institute of Health Stroke Scale (NIHSS) ≥ 4 points;（5）.Glasgow coma standard (GCS)>7 points;（6）.No serious disability before admission, and modified Rankin Scale (mRS) ≤ 3;（7）. The patient himself or his immediate family members signed the informed consent form.

Exclusion Criteria:

- (1) Cerebral hemorrhage or subarachnoid hemorrhage; (2) Cerebellar and brainstem infarction (including lacunar infarction); (3) Cerebral herniation is formed upon admission; (4) Patients with severe heart, lung, liver, and kidney diseases; (5) Severe upper gastrointestinal bleeding occurred after the onset; (6) The patient has participated in other clinical trials within the past 3 months; (7) Patients with mental illness, or those with severe cognitive impairment (MMSE score ≤9 points) (8) Those with a pacemaker, a metal foreign body at the treatment site, or a severe bleeding tendency.

(9) The investigator believes that other diseases accompanied by the patient may interfere with the correct evaluation of neurological function, or participating in this trial may cause other complications in the patient.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
NIHSS SCALE | 4 weeks
  NIHSS was created by the National Institutes of Health and has good reliability and validity. It has been widely used to evaluate the severity and prognosis of stroke. The scale consists of consciousness, gaze, vision, facial paralysis, movement, sensation, mutual aid, language, neglect and other items, with a maximum score of 33 points.

SECONDARY OUTCOMES:
Stroke Scale of Traditional Chinese Medicine, SSTCM | 4 weeks
  SSTCM mainly includes two parts: TCM symptoms and tongue and pulse conditions. There are a total of 24 symptoms of TCM symptoms. According to their severity and impact on daily life, each item is scored into 4 grades, with 0 points for normal, 1 point for mild, 2 points for moderate, and 3 points for severe. Tongue and pulse conditions are only recorded and not scored. The total score is the sum of the scores of TCM symptoms in Part 1. The higher the score, the more severe the symptoms and the greater the impact on life.
modified Barthel Index, mBI | 4 weeks
  The mBI scale is mainly used to evaluate the self-care ability of patients in daily life. It can be summarized as the patients' independent activities in an indoor environment, such as eating, dressing, and toileting, with a total of ten items. The score of each item is divided into 5 levels, the lowest is 1 and the highest is 5. The higher the level, the greater the independence, and the total score is 100 points.

OTHER OUTCOMES:
CRP | baseline ,4 weeks
  acute ischemic biomarker
BDNF | baseline ,4 weeks
  acute ischemic biomarker
MMP-9 | baseline ,4 weeks
  acute ischemic biomarker

CONTACTS AND LOCATIONS:
Overall Officials: jian pei, doctor, Study Director — Longhua Hospital

IPD SHARING:
Plan to Share IPD: Undecided